CLINICAL TRIAL: NCT03220646
Title: A Phase 2 Study of Abemaciclib in Patients With Recurrent Primary Brain Tumors
Brief Title: Abemaciclib (LY2835219) in Patients With Recurrent Primary Brain Tumors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 17-261
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Brain Tumor
Keywords: Abemaciclib (LY2835219); meningioma; Astrocytoma; ependymoma; Oligodendroglioma; CNS lymphoma; 17-261
MeSH Terms: conditions — Brain Neoplasms; Meningioma; Astrocytoma; Ependymoma; Oligodendroglioma | interventions — abemaciclib

STUDY DESIGN:
Intervention Model Description: This is an open-label, non-randomized, phase II trial of single-agent abemaciclib administered at previously defined MTD/RP2D in three cohorts of patients with primary brain tumors.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- A:recurrent IDH wildtype RB1 intact grade II and III gliomas (Experimental): The main study cohort will consist of patients with recurrent IDH wildtype, RB1 wildtype, WHO grade II and III gliomas that have failed previous therapy. This arm is currently on hold.
  Interventions: Drug: abemaciclib
- B:Recurrent glioma any grade (Experimental): Ten patients who require standard of care cytoreductive surgery for recurrent astrocytoma, oligodendroglioma, or glioblastoma, will be offered pre-surgical abemaciclib and then resume the drug following recovery from surgery, continuing until disease progression or unacceptable toxicity analogous to the non-surgical patients in cohort A and C. This arm is closed to accrual.
  Interventions: Drug: abemaciclib
- C:All other recurrent brain tumors (Experimental): This is an exploratory cohort including patients with recurrent IDH mutant glioma, meningioma, recurrent ependymoma, and recurrent PCNSL,and other primary brain tumors.
  Interventions: Drug: abemaciclib

INTERVENTIONS:
Drug: abemaciclib — abemaciclib 200mg PO q12 hours (+/- 2 hours) on days 1-28 of each 28 day cycle.
  Arms: A:recurrent IDH wildtype RB1 intact grade II and III gliomas; C:All other recurrent brain tumors
Drug: abemaciclib — 200mg PO q12 hours (+/- 2 hours) for 4-7 days prior to surgery. Upon recovery from surgery, patients will resume abemaciclib at the same dose and schedule as cohorts A and C.
  Arms: B:Recurrent glioma any grade

SUMMARY:
The purpose of this study is to test any good and bad effects of a study drug called abemaciclib (LY2835219) in patients with recurrent brain tumors.

ELIGIBILITY:
Inclusion Criteria:

Cohort A specific inclusion:

* Histologically confirmed IDHwt, RB intact, grade II or III glioma that has recurred after first line therapy (consisting of at least maximum feasible surgical resection and radiation therapy). There is no limit on the number of prior therapies or types of therapies patients can have received.
* Measurable disease on imaging (1cm) or measurable non-enhancing tumor.
* At least 12 weeks elapsed since prior radiotherapy

Cohort B specific inclusion:

* Patients with histologically confirmed glioma of any grade (II-IV) who are planned for a standard of care surgical debulking/resection and for whom participation in this study would not cause a medically unacceptable delay in surgery.
* Patients must have relapsed/progressed following therapy (consisting of at least maximum feasible surgical resection and radiation therapy).

Cohort C specific Inclusion:

* Histologically confirmed IDH mutant glioma, meningioma, schwanomma, PCNSL, ependymoma, or other Primary Brain Tumors that have recurred despite previous standard of care therapy. Because this cohort is, in part, meant to allow patients access to therapy who might not otherwise be eligible for other clinical trials - deviations from standard of care treatment or histological confirmation can be presented to and approved by the Principal Investigator for inclusion in the study.
* Histologically confirmed PCNSL that has recurred after prior methotrexate-based chemotherapy or for whom methotrexate-based chemotherapy is deemed medically not in the patient's best interest.

Glioma patients:

* Standard of care next generation sequencing via a CLIA certified platform must be available, or planned and at a minimum include IDH, and RB status.

All cohorts:

* Patients must provide written informed consent prior to any screening procedures.
* Age 18 years or older.
* KPS ≥ 60
* Willing and able to comply with scheduled visits, treatment plan and laboratory tests
* Patient is able to swallow and retain oral medication
* Required baseline laboratory status:

  * Hemoglobin > 8 g/dL (SI Units: 80 g/L). Patients may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Initial treatment must not begin earlier than the day after the erythrocyte transfusion.
  * Platelet count ≥ 100 x 10^9/L
  * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L without growth factor support
  * Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
  * AST/SGOT and/or ALT/SGPT ≤ 3 x ULN
  * Serum Creatinine ≤ 1.5 x ULN
* Stable dose of corticosteroids for > 5 days prior to baseline MRI
* Before starting study treatment, patients must have recovered from toxic effects of prior therapies (except for residual alopecia or Grade 2 peripheral neuropathy) and at least 3 weeks must have elapsed since any prior signaling pathway modulators, (e.g., EGFR, FGFR, or other tyrosine kinase inhibitors), at least 3 weeks must have elapsed since temozolomide, 4 weeks must have elapsed since carboplatin or cisplatin, and at least 6 weeks from nitrosoureas (e.g., BCNU, CCNU). In general, at least 4 weeks must have elapsed from any other anticancer drug therapy (e.g. bevacizumab).
* Patients must be able to undergo contrast enhanced MRI scans (or contrast enhanced CT scans for patients unable to tolerate MRI).
* Patients must have shown unequivocal evidence for tumor progression by MRI (or CT for patients who cannot tolerate MRI) in comparison to a prior scan. The same type of scan, i.e., MRI (or CT for patients who cannot undergo MRI) must be used throughout the period of protocol treatment for tumor measurement.
* Life expectancy of greater than 8 weeks
* If a female of childbearing potential, must have a negative serum pregnancy test within 7 days of the first dose of abemaciclib and agree to use a medically approved contraceptive method during the treatment period and for 3 months following the last dose of abemaciclib. If a male, agree to use a reliable method of birth control and to not donate sperm during the treatment period and for at least 3 months following the last dose of abemaciclib. Contraceptive methods may include an intrauterine device [IUD] or barrier method. If condoms are used as a barrier method, a spermicidal agent should be added as a double barrier protection.

Note: Cases of pregnancy that occur during maternal exposures to abemaciclib should be reported. If a patient or spouse/partner is determined to be pregnant following abemaciclib initiation, she must discontinue treatment immediately. Data on fetal outcome and breast-feeding are collected for regulatory reporting and drug safety evaluation.

* Women must agree not to breast feed while on abemaciclib treatment and for at least three months following the last dose of study therapy.

Exclusion Criteria:

* No limit on number of prior therapies
* Evidence of significant intracranial hemorrhage
* No other investigational or standard anti-tumor therapy allowed
* Patients must not have a known history of allergic reactions attributed to compounds of similar chemical or biologic composition.
* Patients must not have a serious preexisting medical condition(s) or uncontrolled intercurrent illness that would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea) or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients who have a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological original (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions. This applies only to patients who have a documented history of HIV; HIV testing is not otherwise required.
* Have an active systemic fungal and/or known viral infection (for example, human immunodeficiency virus antibodies, hepatitis B surface antigen, or hepatitis C antibodies)
* Patients must not be on EIAEDs
* Females who are pregnant or lactating
* Must abstain from grapefruit juice
* Patients must not have other active concurrent malignancy
* Concurrent treatment on another clinical trial. Supportive care trials or non-therapeutic trials (i.e. Quality of life) are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-07-13 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
radiographic response rate | 6 months
  MRI (or CT) scan by RANO criteria.
progression free survival (PFS) | 6 months
  will be estimated by the Kaplan Meier method

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kaley, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Hartford Healthcare Cancer Institute @ Hartford Hospital (Data collection only), Hartford, Connecticut
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Lehigh Valley Health Network, Allentown, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kaley TJ, Grommes C, Coffee E, Young RJ, Morrison T, Daher A, Schaff LR, Deng Y, Nandakumar S, Diamond EL, DeAngelis LM, Panageas KS, Gavrilovic I, Lin A, Pentsova E, Stone J, Santomasso BD, Piotrowski AF, Nair S, Schultz N, Reiner AS, Mellinghoff IK. Multicenter basket trial for Central Nervous System tumors identifies activity of the CDK4/6 inhibitor abemaciclib in recurrent meningioma. Neuro Oncol. 2025 Aug 16:noaf184. doi: 10.1093/neuonc/noaf184. Online ahead of print. PMID 40842355
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm